CLINICAL TRIAL: NCT01821456
Title: The Cologne Cohort of Neutropenic Patients (CoCoNut) - a Non-interventional Cohort Study Assessing Risk Factors, Interventions, and Outcome of Immunosuppressed Patients With or Without Opportunistic Infections
Brief Title: Cologne Cohort of Neutropenic Patients (CoCoNut)
Acronym: CoCoNut
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Sponsor
Other Study IDs: !SZINF2; !!SZINF2 (Other: University Hospital of Cologne)
Record Dates: First submitted 2013-03-19; First posted 2013-04-01 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-03

CONDITIONS: Hematological Malignancies; Cancer; Chemotherapy; Neutropenia; Immunosuppression
Keywords: hematological malignancies; cancer; chemotherapy; anti-infectives; treatment; outcome
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms; Neutropenia | interventions — Anti-Infective Agents; Antifungal Agents; Antiviral Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Antiinfectives: To analyze the efficacy of antiinfectives at high risk patients
  Interventions: Drug: Antiinfectives

INTERVENTIONS:
Drug: Antiinfectives — To analyze to efficacy of (novel) drug therapies
  Other Names: Antifungals, Antibacterials, Antivirals

SUMMARY:
The Cologne Cohort of Neutropenic Patients (CoCoNut) is a non-interventional cohort study assessing risk factors, interventions, and outcome of immunosuppressed patients with or without opportunistic infections.

DETAILED DESCRIPTION:
This prospective cohort was established with the aim of a comprehensive data collection of all patients developing neutropenia after receiving chemotherapy for any kind of malignant disease, treated in the University Hospital of Cologne.

ELIGIBILITY:
Inclusion Criteria:

* immunosuppressed patients

Exclusion Criteria:

* none

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients developing neutropenia after receiving chemotherapy for any kind of malignant disease, treated in the University Hospital of Cologne
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 1995-01; Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Long-term survival of hematology and oncology patients following neutropenia | 2 years following last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Vehreschild JJ, Ruping MJ, Wisplinghoff H, Farowski F, Steinbach A, Sims R, Stollorz A, Kreuzer KA, Hallek M, Bangard C, Cornely OA. Clinical effectiveness of posaconazole prophylaxis in patients with acute myelogenous leukaemia (AML): a 6 year experience of the Cologne AML cohort. J Antimicrob Chemother. 2010 Jul;65(7):1466-71. doi: 10.1093/jac/dkq121. Epub 2010 Apr 21. PMID 20410061
- [Derived] Vehreschild MJ, von Bergwelt-Baildon M, Tran L, Shimabukuro-Vornhagen A, Wisplinghoff H, Bangard C, Cornely OA, Vehreschild JJ. Feasibility and effectiveness of posaconazole prophylaxis in combination with micafungin bridging for patients undergoing allogeneic stem cell transplantation: a 6-yr analysis from the cologne cohort for neutropenic patients. Eur J Haematol. 2014 Nov;93(5):400-6. doi: 10.1111/ejh.12368. Epub 2014 May 26. PMID 24798021
- [Derived] Vehreschild MJ, Weitershagen D, Biehl LM, Tacke D, Waldschmidt D, Tox U, Wisplinghoff H, Von Bergwelt-Baildon M, Cornely OA, Vehreschild JJ. Clostridium difficile infection in patients with acute myelogenous leukemia and in patients undergoing allogeneic stem cell transplantation: epidemiology and risk factor analysis. Biol Blood Marrow Transplant. 2014 Jun;20(6):823-8. doi: 10.1016/j.bbmt.2014.02.022. Epub 2014 Mar 6. PMID 24607558